CLINICAL TRIAL: NCT03780075
Title: Lu177-EB-PSMA617 Prostate-Specific Membrane Antigen Inhibitor Therapy in Patients With Castration-Resistant Prostate Cancer
Brief Title: Lu177-EB-PSMA617 Radionuclide Treatment in Patients With Metastatic Castration-resistant Prostate Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PekingUMCH-NM019
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Metastatic Castration-resistant Prostate Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1.11GBq of 177Lu-EB-PSMA-617 (Experimental): The patients were intravenously injected with the dose about 1.11GBq (30 mCi) of 177Lu-EB-PSMA617 and underwent 68Ga-PSMA PET/CT scans before and after the treatment.
  Interventions: Drug: 1.11GBq of 177Lu-EB-PSMA-617
- 2.00 GBq of 177Lu-EB-PSMA-617 (Experimental): The patients were intravenously injected with the dose about 2.00 GBq (54 mCi) of 177Lu-EB-PSMA-617 and underwent 68Ga-PSMA PET/CT scans before and after the treatment.
  Interventions: Drug: 2.00 GBq of 177Lu-EB-PSMA-617
- 3.70GBq of 177Lu-EB-PSMA-617 (Experimental): The patients were intravenously injected with the dose about 3.70GBq (100 mCi) of 177Lu-EB-PSMA617 and underwent 68Ga-PSMA PET/CT scans before and after the treatment.
  Interventions: Drug: 3.70GBq of 177Lu-EB-PSMA-617

INTERVENTIONS:
Drug: 1.11GBq of 177Lu-EB-PSMA-617 — Patients were intravenous injected with the dose about 1.11GBq (30 mCi) of 177Lu-EB-PSMA-617 every 8 weeks (±1 week) for a maximum of 3 cycles.
  Arms: 1.11GBq of 177Lu-EB-PSMA-617
Drug: 2.00 GBq of 177Lu-EB-PSMA-617 — Patients were intravenous injected with the dose about 2.00 GBq (54 mCi) of 177Lu-EB-PSMA-617 every 8 weeks (±1 week) for a maximum of 3 cycles.
  Arms: 2.00 GBq of 177Lu-EB-PSMA-617
Drug: 3.70GBq of 177Lu-EB-PSMA-617 — Patients were intravenous injected with the dose about 3.70GBq (100 mCi) of 177Lu-EB-PSMA-617 every 8 weeks (±1 week) for a maximum of 3 cycles.
  Arms: 3.70GBq of 177Lu-EB-PSMA-617

SUMMARY:
In prior studies, the investigators synthesized 177Lu-EB-PSMA-617 by conjugating a truncated Evans Blue (EB) molecule and DOTA chelator onto PSMA-617 and labeled it with 177Lu to increase the tumor accumulation and retention for radioligand therapy，and then the investigators evaluated the dosimetry of 177Lu-EB-PSMA-617 and response to single low-dose treatment in patients with metastatic castration-resistant prostate cancer(mCRPC). This study was performed to evaluate the safety and therapy response to 177Lu-EB-PSMA-617 in patients with mCRPC.

This is an open-label, randomized study. Different groups with doses of 1.11GBq (30 mCi), 2.00 GBq (54 mCi) and 3.7GBq (100 mCi)of 177Lu-EB -PSMA617 will be injected intravenously. All patients will undergo 68Ga-PSMA PET/CT scans before and after the treatment.

DETAILED DESCRIPTION:
Prostate cancer (PC) is the second most common cancer worldwide in men, with persistently high numbers dying from this disease. Recent studies have demonstrated the possibility of 177Lu-PSMA-617 therapy as a viable treatment option in mCRPC. To increase tumor accumulation and retention for radioligand therapy, and reduce dosage of 177Lu, the investigators conjugated a truncated Evans blue (EB) molecule and DOTA chelator onto PSMA-617 (EB-PSMA-617) and label it with 177Lu.

The study is open-label and patients will be divided into three groups and monitored throughout the 6 to 10-month treatment period for survival, disease progression, and adverse events to evaluate the safety and therapy response to the 177Lu-EB-PSMA-617.

ELIGIBILITY:
Inclusion Criteria:

* progressive metastatic castration-resistant prostate cancer that did not respond to androgen-suppression therapy and/or systemic chemotherapy.
* Distant metastases with high PSMA expression confirmed by 68Ga-PSMA PET/CT within one week before the injection of 177Lu-EB-PSMA-617.

Exclusion Criteria:

* a serum creatinine level of more than 150μmol per liter,
* a hemoglobin level of less than 10.0 g/dl,
* a white-cell count of less than 4.0× 109/L,
* a platelet count of less than 100 × 109/L,
* a total bilirubin level of more than 3 times the upper limit of the normal range,
* a serum albumin level of more than 3.0 g per deciliter,
* cardiac insufficiency including carcinoid heart valve disease,
* a severe allergy or hypersensitivity to radiographic contrast material,
* claustrophobia, and pregnancy or breastfeeding.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-04-15 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change of the PSA and standardized uptake value of 68Ga-PSMA before and after the treatment in mCRPC | 1 year
  The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake in lesions will be measured.

SECONDARY OUTCOMES:
Adverse events collection | patients will be monitored throughout the whole treatment period. Patients will be followed up every 3 month until 1 year for a long-term follow-up period.
  Adverse events after the treatment of patients will be followed and assessed

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD,PHD, Study Chair — Peking Union Medical College Hospital, Chinese Academy of Medical Science
Locations (1):
- Peking Union Medical College Hospital, Beijing, China